CLINICAL TRIAL: NCT06009484
Title: Incidence of Venous Thrombotic Event After Curative Colon Cancer Surgery in an Enhanced Recovery After Surgery Program
Brief Title: VTE Incidence After Curative Colon Cancer Surgery in an ERAS Program
Status: Completed | Type: Observational
Sponsor: Nordsjaellands Hospital (Other)
Collaborators: Bispebjerg Hospital (Other); Herlev and Gentofte Hospital (Other); Hvidovre University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: VTE-1
Record Dates: First submitted 2023-08-18; First posted 2023-08-24 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Deep Vein Thrombosis, Pulmonary Embolus; Colon Cancer
Keywords: Prolonged thromboembolic prophylaxis
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism; Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 60 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Colon resection — Colon cancer resection

SUMMARY:
Based on data on a cohort of 2,141 patients undergoing elective colonic cancer resection in an ERAS program, the incidence of postoperative thromboembolic events is estimated in patients no receiving prolonged thromboembolic prophylaxis.

DETAILED DESCRIPTION:
The Copenhagen cOmplete Mesocolic Excision Study (COMES) database contains comprehensive data on preoperative, intraoperative, postoperative and tumor related variable on patients undergoing elective colonic cancer resection at four public university clinics providing all colorectal cancer treatment for the 1.8 million residents of the Capital Region of Denmark during the period 2014-2017.

None of these hospitals had implemented prolonged thromboembolic prophylaxis after discharge.

The medical records were reviewed with focusing on VTE prophylaxis, ongoing preoperative and postoperative anticoagulant treatment, the length of hospital stay (LOS), and readmission to ensure high data validity.

ELIGIBILITY:
Inclusion Criteria:

* elective macroradical resection for UICC Stage I-III colonic adenocarcinoma

Exclusion Criteria:

* concomitant rectum resection
* soly appendix carcinoma
* diagnosed with pulmonary embolism or deep venous thrombosis before primary discharge
* dying before discharge from the hospital or discharged at postoperative day 28 or later
* treatment with vitamin K antagonists, heparin or new oral anticoagulants before or after surgery
* VTE less than 3 months before the colon resection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective macroradical resection for UICC Stage I-III colonic adenocarcinoma in the Capital Region of Denmark between January 1, 2014, and December 31, 2017. The database does not include acute cases, cases of metachronous colorectal cancers or rectal cancers without synchronous colonic adenocarcinoma.
Sampling Method: Non-Probability Sample
Enrollment: 2141 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-03-15 (Actual)

PRIMARY OUTCOMES:
Postoperative venous thromboembolic event | 60 days
  Deep venous thrombosis or pulmonary embolism

CONTACTS AND LOCATIONS:
Overall Officials: Claus A Bertelsen, Ph.D., Study Chair — Copenhagen University Hospital - North Zealand

IPD SHARING:
Plan to Share IPD: No